CLINICAL TRIAL: NCT02856685
Title: A Phase 1/2 Study of Mitoxantrone Hydrochloride Liposome Infusion in Patients With Non-Hodgkin's Lymphoma
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Infusion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-AB-NHL-01
Record Dates: First submitted 2016-08-01; First posted 2016-08-05 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PLM60 (Experimental): Mitoxantrone Hydrochloride Liposome
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — Mitoxantrone Hydrochloride Liposome will be administered via IV infusion over 60 minutes once at the beginning (Day 1) of each 28-day cycle
  Other Names: PLM60

SUMMARY:
This is a Phase 1/2, open-label, multicenter study.

DETAILED DESCRIPTION:
The Phase 1 part of this study is designed to identify the MTD and RP2D, and to characterize the safety, tolerability, and PK. The Phase 1 part of the study will include 2 parts: dose escalation and dose expansion.

After confirmation of the RP2D in the expansion part of Phase 1, enrolment into the Phase 2 part of the study will begin. The primary objective of the Phase 2 part of the study is to evaluate the efficacy of the investigational drug when administered to patients with relapsed or refractory NHL.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to study-related procedures
* Patients with histologically confirmed, relapsed or refractory NHL after treatment with standard regimens. Patients with both intermediate and aggressive subtypes (for example, diffuse large B-cell lymphoma, mantle cell lymphoma, peripheral T-cell lymphoma, anaplastic large-cell lymphoma) and indolent subtypes that require treatment (for example, follicular lymphoma, small lymphocytic lymphoma) will be enrolled into the Phase 1 part of the study; Patients with indolent types of NHL must have been assessed as needing further treatment by the Investigator, based on the presence of lymphoma-related symptoms or the presence of significant tumor burden;(Phase 1)
* Adult patients with histologically confirmed relapsed or refractory aggressive NHL (including diffuse large B-cell lymphoma, peripheral T-cell lymphoma, and natural killer cell lymphoma) who were treated with standard regimens and for whom there is no known effective therapy;(Phase 2)
* > 4 weeks since last cycle of chemotherapy prior to the study drug administration;
* Recovered from all toxicity from prior chemotherapy at Investigator's discretion;
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance score of 0-2;
* Patients who have sufficient baseline organ function and whose laboratory data meet the following criteria at enrolment: Absolute neutrophil count ≥ 1.5 x 109/L; Platelets ≥ 75 x 109/L; Hemoglobin ≥ 90 g/L (unless bone marrow involvement is present); Liver function: Serum bilirubin ≤ 1.2 x upper limit of normal (ULN), Aspartate aminotransferase and alanine aminotransferase ≤ 3 x ULN without liver metastases or ≤ 5 x ULN if the patient has documented liver metastases; International normalization ratio < 1.3 if the patient is not on anticoagulants or < 3 if the patient is on anticoagulants o Serum creatinine ≤ 1.5 mg/dL or estimated glomerular filtration rate > 40 mL/min/m2;
* Left ventricular ejection fraction (LVEF) > 50%;
* Life expectancy ≥ 12 weeks;
* Women of childbearing potential must have a negative pregnancy test prior to study entry, and agree to use adequate contraception from study entry through at least 3 months after the last dose of study drug. Adequate methods of contraception for patient or partner include vasectomized partner (at least 6 months prior to dosing); intrauterine device; condom with spermicidal gel, foam, cream, film, or suppository; diaphragm with spermicidal gel, foam, cream, film, or suppository; or cervical cap with spermicidal gel, foam, cream, film, or suppository.A female patient of non-childbearing potential must have had at least 12 continuous months of natural (spontaneous) amenorrhea, follicle-stimulating hormone level > 40 mIU/mL at Screening, or have had surgical bilateral oophorectomy or a hysterectomy > 6 weeks prior to Screening;
* A male patient must agree to use adequate contraception (male condom with spermicide; sterile sexual partner; or female sexual partner who uses an intrauterine device with spermicide, a female condom with spermicide, a contraceptive sponge with spermicide, an intravaginal system, a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives) from study entry through at least 3 months after the last dose of study drug;
* Involved lymph nodes or masses should be measurable in at least 2 perpendicular dimensions and be > 1.5 cm in the longest of the perpendicular dimensions (based on Cheson et al 2014) (Additional Inclusion Criteria for Phase 2);
* Agree to undergo pretreatment bone marrow biopsy and post-treatment bone marrow biopsy when required to confirm response (Additional Inclusion Criteria for Phase 2).

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Patients with a history of allergy to anthracyclines or liposomal drugs;
* Prior treatment with mitoxantrone;
* Treatment with doxorubicin with a total cumulative dose > 300 mg/m2, or epirubicin with the total cumulative dose > 500 mg/m2;
* Investigational treatment within 4 weeks of the start of PLM60;
* Systemic chemotherapy within 4 weeks of the start of PLM60;
* Radiotherapy (≥25 % of bone marrow) within 4 weeks of the start of PLM60;
* Radio-/toxin-immunoconjugates within 42 days of the start of PLM60;
* Prior allogeneic stem cell transplantation;
* Known central nervous system involvement by NHL;
* Patients who have the following types of cardiac impairment at the time of enrolment: New York Heart Association class III or IV heart disease; Uncontrolled angina, congestive heart failure, or myocardial infarction within 6 months prior to enrolment; An LVEF by echocardiogram or multi-gated acquisition (MUGA) scan < 50%; QT interval prolongation (> 450 ms in males, > 470 ms in females);
* A past history of cardiac disease caused by anthracyclines;
* History of malignancy other than NHL in the past 3 years prior to enrolment, except for adequately treated non-melanoma skin cancer or in situ cervical cancer;
* Patients with evidence of an active infection including the following: Patients being treated with antibiotics for an active infection at the time of enrolment; Patients who have evidence of active hepatitis C or chronic active hepatitis B; Patients who have a known diagnosis of human immunodeficiency virus (HIV) infection/ acquired immunodeficiency syndrome (AIDS);
* Other severe or poorly controlled illness or circumstance that would interfere with evaluation of key study endpoints or which would put the patient at risk from participating in the study in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)(Phase 1) | 28 day cycle of therapy
  Phase 1 -MTD defined as the highest dose level in which 6 patients have been treated with less than 2 instances of dose limiting toxicity (DLT). Dose limiting toxicity is based on adverse events and includes unacceptable hematologic toxicity, unacceptable non-hematologic toxicity, and laboratory abnormalities of Grade 4 or higher.
Objective response rate (ORR; complete response + partial response [CR + PR])(Phase 2) | Approximately 2 years
  Tumor response and progression will be evaluated every 8 weeks according to the Lugano Classification (Cheson et al 2014).

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of PLM60 | Approximately 1 years

OTHER OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time zero to the time point of t (AUC0-t) | Approximately 1 years
Area under the plasma concentration-time curve (AUC) from time zero to infinity (AUC0-∞) | Approximately 1 years
Apparent terminal phase elimination rate constant (λz) | Approximately 1 years
Apparent terminal elimination half-life (T½β) | Approximately 1 years
Apparent volume of distribution (V) | Approximately 1 years
Total clearance (CL/F) | Approximately 1 years
Distribution volume (Vd/F) | Approximately 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Nashat Y Gabrail, M.D., Principal Investigator — Gabrail Cancer Center Research
Locations (1):
- Gabrail Cancer Center Research, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes